CLINICAL TRIAL: NCT06573346
Title: Investigation of the Effect of Cervical Stabilization Exercises on Bruxism and Sleep Quality
Brief Title: Cervical Stabilization Exercises on Bruxism and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Emine Nur Demircan, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cervical stabilization
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-08

CONDITIONS: Bruxism; Sleep Quality; Cervical Stabilization Exercise
MeSH Terms: conditions — Bruxism; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Other: Cervical spinal stabilization exercise
- Experimental group (Experimental)
  Interventions: Other: Cervical spinal stabilization exercise

INTERVENTIONS:
Other: Cervical spinal stabilization exercise — The cervical region is one of the most affected regions of the musculoskeletal system due to the intensive proprioceptors. Studies have shown that many position sense proprioceptors are over the deep group cervical muscles such as longus colitis and longus capitis. The deep group cervical muscles, which perform a dynamic ligament function, have an important role in maintaining the stability of the spine as well as the proprioceptive sense. In particular, proprioceptive receptors, which are commonly found in the deep suboccipital muscles; There are cervical and reflex connections with vestibular, visual and postural control systems.

SUMMARY:
Bruxism and temporomandibular joint dysfunction are common conditions today. The applications in the treatment of these disorders are limited. When the literature is examined, it has been determined that cervical stabilization exercises, which are frequently applied in physical therapy clinics for neck problems, have not been applied to bruxism before. For this reason, in this study, we will examine the effects of cervical stabilization exercises targeting deep cervical muscles on bruxism.

DETAILED DESCRIPTION:
Bruxism is the grinding or clenching of teeth, which is characterized by the fixed or forward movement of the mandible that occurs repeatedly during the day, including muscles such as the masseter and temporal muscles. Correct determination of the etiology plays a key role in the treatment of bruxism. There are many suggestions in the literature for the treatment of bruxism. The most preferred of these are: providing training for the person to quit harmful habits, physiotherapy applications for muscle relaxation, botox applications, drug treatments, giving the patient an occlusal splint, etc. Since bruxism is a functional problem of muscular origin, it is possible to talk about muscle-oriented exercise applications in its treatment. As a result of studies in which exercises are frequently prescribed for the chewing muscles and temporomandibular muscles, it has been determined that bruxism symptoms are relieved and functional gains are achieved. It has also been stated that muscle pain and activity, mouth opening, oral health, anxiety, stress, depression and head posture can be improved in individuals with bruxism with physiotherapy approaches. When the literature is examined; There are studies investigating the effects of physiotherapy applications in bruxism. In addition, although it is known that the neck region is affected in bruxism, causing the head to tilt forward and increased muscle activation in the neck region, no study has been found investigating the effects of specific cervical region stabilization exercises. This study was planned considering the effects of cervical stabilization exercises on correcting cervical posture and providing muscle activation balance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with full dentition including 2nd molars
* Patients without facial asymmetry

Exclusion Criteria:

* Patients with systemic and/or neuromuscular diseases
* Patients with orofacial pain not caused by bruxism
* History of temporomandibular joint (TMJ) surgery or injection
* Use of any medical drugs affecting the muscular system
* Patients with developmental deformities or a history of surgery in the maxillofacial region (facial trauma history, resection history, etc.)
* TMJ pathologies (major condylar changes seen on panoramic radiographs)
* History of radiotherapy and/or chemotherapy
* Ongoing orthodontic treatment
* Use of removable prosthesis
* Inflammatory connective tissue diseases
* Pregnancy
* Obstructive sleep apnea
* Local skin infection over the myofascial area
* Patients who have undergone root canal treatment
* Reluctance to take responsibility for the work

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Muscle Activation Evaluation | At baseline, after 6 weeks of treatment, 4 weeks after the end of treatment
  Participants' Masseter, Temporal and Trapezius muscle activation will be evaluated with Superficial Electromyography. (Number of Participants estimated 28 individuals)
Tongue Pressure Evaluation | At baseline, after 6 weeks of treatment, 4 weeks after the end of treatment
  Tongue pressure will be done by oral muscle measurement. (Number of Participants estimated 28 individuals)
Evaluation of Sleep Quality | At baseline, after 6 weeks of treatment, 4 weeks after the end of treatment
  Since bruxism affects the sleep quality of patients, the Pittsburg Sleep Quality Index will be used to evaluate sleep quality. (Number of Participants estimated 28 individuals)

SECONDARY OUTCOMES:
Mouth Opening Evaluation | At baseline, after 6 weeks of treatment, 4 weeks after the end of treatment
  The amount of mouth opening will be evaluated by adding the vertical coverage amounts of the lower and upper incisors to the distance between the incisal edges of the lower and upper incisors at maximum mouth opening, using a ruler, for pre-treatment, post-treatment and 1 month later follow-up purposes. (Number of Participants estimated 28 individuals)
Tongue Range of Motion Ratio Assessment | At baseline, after 6 weeks of treatment, 4 weeks after the end of treatment
  In the functional tongue tie classification published by Ferrés-Amat et al., the mouth opening with tongue tip to maxillary incisive papillae at roof of mouth (MOTTIP) and the maximum interincisal mouth opening (MIO) ratio (MOTTIP/MIO ratio is defined as "Tongue range of motion ratio - TRMR") will be used to measure functional tongue limitation. In this classification system, it is stated as Grade 1: tongue range of motion ratio >% 80, Grade 2: 50-80, Grade 3: <% 50, Grade 4: <% 25. (Number of Participants estimated 28 individuals)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kent University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lobbezoo F, Ahlberg J, Glaros AG, Kato T, Koyano K, Lavigne GJ, de Leeuw R, Manfredini D, Svensson P, Winocur E. Bruxism defined and graded: an international consensus. J Oral Rehabil. 2013 Jan;40(1):2-4. doi: 10.1111/joor.12011. Epub 2012 Nov 4. PMID 23121262
- [Background] Lavigne GJ, Kato T, Kolta A, Sessle BJ. Neurobiological mechanisms involved in sleep bruxism. Crit Rev Oral Biol Med. 2003;14(1):30-46. doi: 10.1177/154411130301400104. PMID 12764018
- [Background] Kato T, Rompre P, Montplaisir JY, Sessle BJ, Lavigne GJ. Sleep bruxism: an oromotor activity secondary to micro-arousal. J Dent Res. 2001 Oct;80(10):1940-4. doi: 10.1177/00220345010800101501. PMID 11706956
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Hirai K, Ikawa T, Shigeta Y, Shigemoto S, Ogawa T. Evaluation of sleep bruxism with a novel designed occlusal splint. J Prosthodont Res. 2017 Jul;61(3):333-343. doi: 10.1016/j.jpor.2016.12.007. Epub 2017 Jan 18. PMID 28109797